CLINICAL TRIAL: NCT07386171
Title: Evaluating Micro-Ultrasound as a Supplemental Imaging Modality for Clinically Significant Prostate Cancer Detection in Men With Negative or Stable Multiparametric MRI on Active Surveillance or at Diagnosis
Brief Title: Micro-Ultrasound for Detecting Clinically Significant Prostate Cancer in Active Surveillance
Acronym: MUS-AS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Rafael Sanchez-Salas, Associate Professor of Urology, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MUHC-MICROUS-AS-2026-01
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Active Surveillance for Prostate Cancer; Imaging Techniques
Keywords: Active Surveillance Prostate Cancer; Prostate Cancer Imaging; Micro-ultrasound; Multiparametric MRI; Clinically significant prostate cancer; Targeted-Systematic biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-arm diagnostic study in which all participants undergo micro-ultrasound assessment. Participants with PRI-MUS ≥3 lesions receive targeted biopsy, and all participants undergo systematic 12-core biopsy during the same session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Micro-Ultrasound Imaging and Biopsy (Experimental): All participants will undergo micro-ultrasound prostate assessment. If a suspicious lesion is identified, targeted biopsy will be performed. All participants will also undergo a 12-core systematic biopsy during the same session.
  Interventions: Diagnostic Test: Micro-Ultrasound (mUS)

INTERVENTIONS:
Diagnostic Test: Micro-Ultrasound (mUS) — High-frequency micro-ultrasound prostate imaging with real-time lesion assessment. Targeted biopsy of suspicious lesions will be performed when present, along with concurrent systematic 12-core biopsy.

SUMMARY:
Active surveillance is a common approach for men with low-risk or favorable intermediate-risk prostate cancer, aimed at avoiding or delaying treatment while closely monitoring the disease. Multiparametric MRI (mpMRI) is widely used to guide diagnosis and follow-up, but it can miss clinically significant prostate cancer and may be limited by access, cost, and variability in interpretation.

Micro-ultrasound is a high-resolution ultrasound technique that may improve real-time detection of suspicious prostate lesions using a standardized scoring system (PRI-MUS). The purpose of this study is to evaluate the diagnostic performance of micro-ultrasound for detecting clinically significant prostate cancer in men with negative or stable mpMRI findings, either at initial diagnosis or during active surveillance follow-up.

Participants will undergo micro-ultrasound assessment of the prostate. Areas considered suspicious on micro-ultrasound may be targeted for biopsy, followed by systematic prostate sampling. Biopsy results will be used as the reference standard to determine whether clinically significant prostate cancer is present.

The study will assess measures such as sensitivity, specificity, and predictive values of micro-ultrasound, as well as procedure-related complications.

DETAILED DESCRIPTION:
Study Rationale This is a prospective, single-arm, two-stage phase II diagnostic study designed to evaluate micro-ultrasound (mUS) as a supplemental imaging modality for the detection of clinically significant prostate cancer (csPCa) in men undergoing active surveillance (AS), or newly diagnosed men eligible for AS, with negative (PI-RADS ≤2) or stable multiparametric MRI (mpMRI) findings.

Active surveillance is widely adopted for men with low-risk and selected favorable intermediate-risk prostate cancer (PCa), aiming to defer or avoid definitive treatment while maintaining oncologic safety through structured monitoring.

mpMRI has become central to risk stratification, patient selection, and follow-up. However, clinically significant disease can be missed despite negative or stable mpMRI findings due to false-negative scans, inter-reader variability, limited access, and cost constraints. These limitations may lead to underdetection of csPCa and potential delays in appropriate treatment. In contrast to mpMRI, mUS can be performed at the point of care during the urology visit, enabling real-time lesion assessment and immediate targeted biopsy without the need to wait for radiology reporting, which may help mitigate MRI-related access delays and workflow bottlenecks.

mUS is a high-frequency ultrasound technology (29 MHz) providing real-time, high-resolution imaging of the prostate, enabling lesion characterization using the Prostate Risk Identification using Micro-Ultrasound (PRI-MUS) scoring system. mUS may detect suspicious features not identified on mpMRI and may therefore improve detection of csPCa, particularly in men with negative or stable mpMRI who are still undergoing biopsy due to clinical triggers or surveillance protocols.

Study Objectives The primary objective of this study is to determine the diagnostic performance of mUS for detecting csPCa in this population, using histopathology as the reference standard.

Secondary objectives include:

* Evaluating positive and negative predictive values of mUS.
* Estimating the incremental detection of csPCa provided by mUS compared with mpMRI alone.
* Evaluating concordance between mpMRI and mUS lesion identification and risk classification.
* Describing biopsy-related adverse events and complications using standardized reporting and grading.

Study Design This is a prospective, single-arm, diagnostic accuracy study incorporating a two-stage phase II design (Simon two-stage design). The study will evaluate whether the detection rate and sensitivity of mUS for csPCa meets a pre-specified threshold that would justify broader implementation or future comparative studies.

The two-stage design allows for early termination for futility if interim results indicate that the diagnostic performance of mUS is insufficient. If the performance targets are met in Stage 1, the study proceeds to Stage 2 to complete the planned sample size and provide more precise estimates of diagnostic accuracy.

Study Population Participants are men aged 45 to 75 years with localized PCa enrolled in AS or newly diagnosed and eligible for AS, who have either negative mpMRI (PI-RADS ≤2) or stable mpMRI findings over time.

Eligibility criteria include features consistent with low-risk or favorable intermediate-risk disease, as determined by prior biopsy results, PSA values, and clinical staging.

Study Procedures All participants will undergo mUS assessment of the prostate according to a standardized imaging protocol. The prostate will be systematically examined, and lesions will be scored using the PRI-MUS risk stratification system. Lesions scored PRI-MUS ≥3 will be considered suspicious and will be targeted for biopsy under micro-ultrasound guidance. Following targeted sampling (when applicable), all participants will undergo systematic prostate biopsy (12-core sampling) during the same procedure session. Targeted and systematic biopsy cores will be analyzed by experienced genitourinary pathologists using standardized reporting. Histopathology will serve as the reference standard for determining the presence or absence of csPCa.

Definition of (csPCa) Clinically significant PCa is defined as Grade Group ≥2 (Gleason score ≥3+4) detected in any biopsy core (targeted or systematic). This definition is aligned with contemporary AS risk thresholds and is intended to capture disease that may warrant treatment escalation or intensified monitoring.

Outcomes

* Primary outcome measures include sensitivity and specificity of mUS for detecting csPCa (Grade Group ≥2). mUS "test positivity" will be defined based on PRI-MUS score thresholds (PRI-MUS ≥3) and/or the presence of a targetable lesion on mUS.
* Secondary outcome measures include positive predictive value (PPV), negative predictive value (NPV), and overall diagnostic accuracy. Incremental csPCa detection attributable to mUS will be assessed by describing csPCa detected in mUS-targeted cores and comparing detection patterns relative to mpMRI findings (negative vs stable findings) and other clinical parameters.

Agreement between mpMRI and mUS lesion identification will be assessed using appropriate concordance metrics (e.g., Cohen's kappa) when applicable.

-Safety outcomes will include biopsy-related adverse events, including infectious complications, urinary retention, bleeding events, pain, and other procedure-related outcomes. Adverse events will be collected prospectively and categorized according to standardized definitions, and clinically relevant complications will be graded using established severity classifications (e.g., Clavien-Dindo).

Statistical Considerations Diagnostic accuracy metrics (sensitivity, specificity, PPV, NPV) will be reported with confidence intervals. The study's two-stage phase II design provides an efficient approach to determining whether mUS demonstrates adequate diagnostic performance for csPCa detection in this clinically important subgroup of men with negative or stable mpMRI findings. Interim analysis will be performed after completion of Stage 1 enrollment and histopathology outcomes, with progression to Stage 2 contingent on meeting the predefined performance threshold.

Clinical Significance This study addresses an unmet need within the AS pathway: improving detection of csPCa in men with negative or stable mpMRI who remain at risk of harboring higher-grade disease. If mUS demonstrates high sensitivity and useful NPV, it may support improved risk stratification, reduce missed csPCa, and optimize biopsy decision-making. The findings may inform future diagnostic strategies and pathway refinement, including how mUS can be integrated with mpMRI in AS and early detection settings.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 45 to 75 years
* Localized prostate cancer on active surveillance or newly diagnosed and eligible for active surveillance
* Negative multiparametric MRI (PI-RADS ≤2) or stable mpMRI findings on surveillance
* Prior prostate biopsy showing Grade Group 1, or Grade Group 2 (Gleason 3+4) with ≤10% pattern 4
* PSA ≤15 ng/mL
* PSA density <0.15 ng/mL/cc
* Clinical stage ≤T2a
* Life expectancy >10 years
* Ability to provide written informed consent and comply with study procedures

Exclusion Criteria:

* Prior definitive treatment for prostate cancer (e.g., radical prostatectomy, radiotherapy)
* Prior prostate surgery that may affect biopsy or imaging interpretation
* Contraindication to prostate biopsy
* Active urinary tract infection or prostatitis
* Inability to tolerate the biopsy procedure or follow study procedures

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants are individuals with a prostate who meet all study inclusion and exclusion criteria.
Enrollment: 90 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Micro-Ultrasound for Clinically Significant Prostate Cancer (Grade Group ≥2) | At the time of the study biopsy procedure (baseline)
  Sensitivity of micro-ultrasound for detecting clinically significant prostate cancer (csPCa), defined as Grade Group ≥2, using histopathology from targeted and systematic biopsy cores as the reference standard.
Specificity of Micro-Ultrasound for Clinically Significant Prostate Cancer (Grade Group ≥2) | At the time of the study biopsy procedure (baseline)
  Specificity of micro-ultrasound for detecting clinically significant prostate cancer (csPCa), defined as Grade Group ≥2, using histopathology from targeted and systematic biopsy cores as the reference standard.

SECONDARY OUTCOMES:
Positive Predictive Value of Micro-Ultrasound for csPCa (Grade Group ≥2) | At the time of the study biopsy procedure (baseline)
  Positive predictive value of micro-ultrasound for detecting clinically significant prostate cancer, defined as Grade Group ≥2, using histopathology as the reference standard.
Negative Predictive Value of Micro-Ultrasound for csPCa (Grade Group ≥2) | At the time of the study biopsy procedure (baseline)
  Negative predictive value of micro-ultrasound for detecting clinically significant prostate cancer (csPCa), defined as Grade Group ≥2, using histopathology as the reference standard.
Overall Diagnostic Accuracy of Micro-Ultrasound for csPCa (Grade Group ≥2) | At the time of the study biopsy procedure (baseline)
  Overall diagnostic accuracy of micro-ultrasound for detecting clinically significant prostate cancer (csPCa), defined as Grade Group ≥2, using histopathology as the reference standard.
Incremental Detection of csPCa Using Micro-Ultrasound Targeted Biopsy | At the time of the study biopsy procedure (baseline)
  Number and proportion of clinically significant prostate cancers (Grade Group ≥2) detected on micro-ultrasound targeted biopsy cores, including csPCa cases that would not have been detected by systematic biopsy alone.
Concordance Between Micro-Ultrasound Findings and mpMRI Findings | At the time of the study biopsy procedure (baseline)
  Agreement between micro-ultrasound and multiparametric MRI findings for lesion identification and risk categorization.

OTHER OUTCOMES:
Biopsy-Related Adverse Events | Up to 30 days post-biopsy
  Incidence and severity of biopsy-related adverse events and complications, graded using standardized criteria (e.g., Clavien-Dindo classification).

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Anidjar, MD, PhD, Study Chair — Jewish General Hospital; Rafael Sanchez-Salas, MD, Principal Investigator — McGill Universiy Health Center // Jewish General Hospital; Rocio Roldan-Testillano, MD, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly to protect participant privacy and confidentiality. De-identified data may be made available upon reasonable request and subject to institutional approvals and applicable ethics requirements.

REFERENCES:
- [Background] Wang L, Lu B, He M, Wang Y, Wang Z, Du L. Prostate Cancer Incidence and Mortality: Global Status and Temporal Trends in 89 Countries From 2000 to 2019. Front Public Health. 2022 Feb 16;10:811044. doi: 10.3389/fpubh.2022.811044. eCollection 2022. PMID 35252092
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Albers P, Wang B, Broomfield S, Medina Martin A, Fung C, Kinnaird A. Micro-ultrasound Versus Magnetic Resonance Imaging in Prostate Cancer Active Surveillance. Eur Urol Open Sci. 2022 Oct 25;46:33-35. doi: 10.1016/j.euros.2022.09.019. eCollection 2022 Dec. PMID 36325366
- [Background] Albers P, Bennett J, Evans M, St Martin E, Wang B, Broomfield S, Martin AM, Tu W, Fung C, Kinnaird A. Micro-ultrasound for the detection of clinically significant prostate cancer in biopsy-naive men with negative MRI. Can Urol Assoc J. 2024 Jun;18(6):208-211. doi: 10.5489/cuaj.8626. PMID 38587980
- [Background] Kinnaird A, Luger F, Cash H, Ghai S, Urdaneta-Salegui LF, Pavlovich CP, Brito J, Shore ND, Struck JP, Schostak M, Harland N, Rodriguez-Socarras M, Brisbane WG, Lughezzani G, Toledano H, Ouertani MS, Macek P, Fung C, Tu W, Gusenleitner A, Gunzel K, Incze PF, George AK, Pereira JG, Jansen R, Renzulli J 2nd, Klotz L; OPTIMUM Investigators. Microultrasonography-Guided vs MRI-Guided Biopsy for Prostate Cancer Diagnosis: The OPTIMUM Randomized Clinical Trial. JAMA. 2025 May 20;333(19):1679-1687. doi: 10.1001/jama.2025.3579. PMID 40121537
- [Background] Basso Dias A, Ghai S. Micro-Ultrasound: Current Role in Prostate Cancer Diagnosis and Future Possibilities. Cancers (Basel). 2023 Feb 17;15(4):1280. doi: 10.3390/cancers15041280. PMID 36831622
- [Background] Scott R, Misser SK, Cioni D, Neri E. PI-RADS v2.1: What has changed and how to report. SA J Radiol. 2021 Jun 1;25(1):2062. doi: 10.4102/sajr.v25i1.2062. eCollection 2021. PMID 34230862
- [Background] Drost FH, Osses D, Nieboer D, Bangma CH, Steyerberg EW, Roobol MJ, Schoots IG. Prostate Magnetic Resonance Imaging, with or Without Magnetic Resonance Imaging-targeted Biopsy, and Systematic Biopsy for Detecting Prostate Cancer: A Cochrane Systematic Review and Meta-analysis. Eur Urol. 2020 Jan;77(1):78-94. doi: 10.1016/j.eururo.2019.06.023. Epub 2019 Jul 18. PMID 31326219
- [Background] Klotz L. Active surveillance in intermediate-risk prostate cancer. BJU Int. 2020 Mar;125(3):346-354. doi: 10.1111/bju.14935. Epub 2020 Jan 16. PMID 31647166
- [Background] Tosoian JJ, Mamawala M, Epstein JI, Landis P, Macura KJ, Simopoulos DN, Carter HB, Gorin MA. Active Surveillance of Grade Group 1 Prostate Cancer: Long-term Outcomes from a Large Prospective Cohort. Eur Urol. 2020 Jun;77(6):675-682. doi: 10.1016/j.eururo.2019.12.017. Epub 2020 Jan 7. PMID 31918957
- [Background] Cornford P, van den Bergh RCN, Briers E, Van den Broeck T, Brunckhorst O, Darraugh J, Eberli D, De Meerleer G, De Santis M, Farolfi A, Gandaglia G, Gillessen S, Grivas N, Henry AM, Lardas M, van Leenders GJLH, Liew M, Linares Espinos E, Oldenburg J, van Oort IM, Oprea-Lager DE, Ploussard G, Roberts MJ, Rouviere O, Schoots IG, Schouten N, Smith EJ, Stranne J, Wiegel T, Willemse PM, Tilki D. EAU-EANM-ESTRO-ESUR-ISUP-SIOG Guidelines on Prostate Cancer-2024 Update. Part I: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2024 Aug;86(2):148-163. doi: 10.1016/j.eururo.2024.03.027. Epub 2024 Apr 13. PMID 38614820
- [Background] Eastham JA, Auffenberg GB, Barocas DA, Chou R, Crispino T, Davis JW, Eggener S, Horwitz EM, Kane CJ, Kirkby E, Lin DW, McBride SM, Morgans AK, Pierorazio PM, Rodrigues G, Wong WW, Boorjian SA. Clinically Localized Prostate Cancer: AUA/ASTRO Guideline, Part I: Introduction, Risk Assessment, Staging, and Risk-Based Management. J Urol. 2022 Jul;208(1):10-18. doi: 10.1097/JU.0000000000002757. Epub 2022 May 10. PMID 35536144